CLINICAL TRIAL: NCT01457898
Title: Effects of Non-invasive Mechanical Ventilation on Hemodynamics and Gas Exchanges Parameters After Cardiac Surgery in Patients With Relative Hypoxemia
Brief Title: Non-invasive Mechanical Ventilation After Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Irmandade Santa Casa de Misericórdia de Porto Alegre (Other)
Collaborators: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Alessandra Preisig, Principal Investigator, Irmandade Santa Casa de Misericórdia de Porto Alegre
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: 1751/07
Record Dates: First submitted 2011-10-19; First posted 2011-10-24 (Estimated); Last update posted 2011-10-25 (Estimated); Status verified 2011-10

CONDITIONS: Heart; Dysfunction Postoperative, Cardiac Surgery
Keywords: Cardiac surgery; Non-invasive ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VPAP II® (Experimental): VPAP II® Group
  Interventions: Device: VPAP II®

INTERVENTIONS:
Device: VPAP II® — VPAP group:inspiratory pressure to generate 6ml/kg of weight and expiratory pressure of 7cmH2O plus oxygen therapy (FIO2=40%) during three hours.
  Other Names: VPAP II -STA (Resmed®)

SUMMARY:
Non-invasive mechanical ventilation (NIV) has been used in hypoxic post-operative cardiac patients but more studies are necessary to clarify its respiratory and hemodynamic effects. Therefore, the investigators objective was to study its effects in the oxygenation index (PaO2/FiO2) and in hemodynamic variables in this group of patients.

DETAILED DESCRIPTION:
* Postoperative cardiac surgery patients having a Swan-Ganz catheter and showing a PaO2/FiO2 between 150 and 300 (with FIO2 0.31), one hour after extubation, were included.
* Then, the patients were randomized into two groups: control and intervention group. Intervention group used NIV with a bi-level positive airway pressure (an inspiratory pressure to generate a tidal volume of 6ml/kg and an expiratory pressure of 7cmH2O) with a FIO2 0.4. Control group used oxygen by Venturi mask(FIO2 0.4) in order to keep a good oxygenation.
* In both groups measurements were done in basal situation, one and three hours after beginning the treatment and one hour after stop the treatment (FiO2 0.31).
* Variables studied included: PaO2/FiO2, PaO2, PaCO2, heart rate (HR), mean arterial pressure (MAP), pulmonary capillary wedge pressure (PCWP) and cardiac output (CO).

ELIGIBILITY:
Inclusion Criteria:

* Oxygenation index (PaO2/FiO2)between 150 and 300 one hour after extubation following cardiac surgery.
* Swan-Ganz catheter

Exclusion Criteria:

* Invasive mechanical ventilation more than 24 hours
* Serious obstructive pulmonary chronic disease (FEV1<40%)

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2008-04; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Oxygenation index (PaO2/FiO2) | 5 hours

SECONDARY OUTCOMES:
Heart rate (HR) | 5 hours
Mean arterial pressure (MAP) | 5 hours
Pulmonary capillary wedge pressure (PCWP) | 5 hours
Cardiac output (CO) | 5 hours

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra P Werlang, MsC, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Santa Casa de Misericórdia de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil